CLINICAL TRIAL: NCT03006978
Title: A Prospective, Single-center, Randomized, Controlled Trial to Evaluate the Safety and Effectiveness of the TearCare System in Adults With Dry Eye Disease TearCare Pilot Study)
Brief Title: A Pilot Study of the TearCare System in Adults With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05429
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TearCare (Experimental): Subjects will receive a 12-minute treatment session with the TearCare System followed by manual expression of the meibomian glands. This procedure will be performed at the Baseline visit.
  Interventions: Device: TearCare
- Warm Compress (Active Comparator): Subjects will apply a warm compress to the eyelids for 5 minutes daily for 4 weeks.
  Interventions: Device: Warm Compress

INTERVENTIONS:
Device: TearCare
  Arms: TearCare
Device: Warm Compress
  Arms: Warm Compress

SUMMARY:
This is a small, pilot study intended to determine the feasibility of this product.

DETAILED DESCRIPTION:
The objective of this study was to evaluate the safety and effectiveness of the TearCare® System in adult patients with clinically significant dry eye disease (DED). This was a prospective, single-center, randomized, parallel-group, clinical trial. Subjects with DED were randomized to either a single TearCare treatment conducted at the clinic or 4 weeks of daily warm compress (WC) therapy. The TearCare procedure consisted of 12 minutes of thermal eyelid treatment immediately followed by manual expression of the meibomian glands. WC therapy consisted of once daily application of the compresses to the eyelids for 5 minutes. Subjects were followed until 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* At Least 18 Years of age
* Reports dry eye symptoms within 3 months of the screening exam with a SPEED score >=6
* Schirmer 1 value of <10 mm in at least one eye or a Tear Breakup time <10 seconds in at least one eye
* Willing to comply with the study, procedures, and follow-up
* Willing and able to provide consent

Exclusion Criteria:

* Any active ocular or peri-ocular infection or inflammation
* Recurrent eye inflammation within the past 3 months
* Ocular surgery, oculoplastic surgery, ocular injury, Ocular Herpes Simplex, or Herpes Zoster
* Ocular surface abnormalities that may affect tear film distribution or treatment
* Abnormal eyelid function in either eye
* Diminished or abnormal facial, periocular, ocular or corneal sensation
* Ocular surface abnormalities such as corneal epithelial defects, ulcers, corneal dystrophies
* Systemic diseases resulting in dry eye (e.g. Sjogren's syndrome)
* Allergies to silicone tissue adhesives
* An absence or fibrosis of the Meibomian glands (e.g. ectodermal dysplasia).
* Unwillingness to abstain for the duration of the study from systemic medication known to cause ocular dryness (e.g. Accutane, antihistamines, etc.)
* Anyone who requires chronic use (i.e. for any portion of the study) of topical ophthalmic antibiotics, steroids, non-steroidal anti-inflammatory medications or who has been on any of these medications within the past 30 days.
* Unwillingness to washout and remain off certain dry eye medications for the duration of the study.
* Participation in another ophthalmic clinical trial within the past 30 days
* Co-existing conditions that could interfere with the assessment of safety or efficacy of treatment (e.g. macular disease, pregnancy, nursing, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Badawi, MD, Principal Investigator — Sight Sciences
Locations (1):
- Central Eye Care, Ltd., Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Badawi D. A novel system, TearCare(R), for the treatment of the signs and symptoms of dry eye disease. Clin Ophthalmol. 2018 Apr 10;12:683-694. doi: 10.2147/OPTH.S160403. eCollection 2018. PMID 29692600

RESULTS

PARTICIPANT FLOW:
Groups:
- TearCare: Subjects will receive a 12-minute treatment session with the TearCare System followed by manual expression of the meibomian glands.
  TearCare
- Warm Compress: Subjects will apply a warm compress to the eyelids for 5 minutes daily for 4 weeks.
  Warm Compress
Period: Overall Study
Arm/Group | TearCare | Warm Compress
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TearCare | Warm Compress | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (11.5) | 66.1 (15.1) | 67.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Tear Breakup Time From Baseline to Month 1
Description: The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit. The change in TBUT was The difference between the mean baseline value and the mean Month 1 value. The TBUT for each eye for a subject was averaged. An increase in TBUT represents an improvement.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TearCare | Warm Compress
Number analyzed (Participants) | 12 | 12
seconds | 11.7 (2.6) | -0.3 (1.1)
Statistical Analysis 1: Comparison: TearCare vs Warm Compress; Test type: Superiority; p < 0.0001, Simple mixed effects linear models

2. Secondary Outcome: Mean Change in Meibomian Gland Score From Baseline to Month 1
Description: Using a Korb Meibomian Gland Evaluator (TearScience), the meibomian gland assessment was conducted by evaluating the consistency of the secretions that were observed upon expression of meibomian glands in the nasal, central, and temporal regions of the lower eyelids. The central, consecutive 5 glands in each region were evaluated. The instrument was held at the eyelid margin for 10-15 seconds, and the secretions were graded on a 0-3 scale for each gland (0=no expression; 1=toothpaste; 2=cloudy; and 3=clear), with a 0-45 score range for each eye. The score for each eye of a subject was averaged. The change from baseline in the Meibomian Gland Score is the difference between the mean baseline value and the mean value at Month 1. A higher score represents an improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare | Warm Compress
Number analyzed (Participants) | 12 | 12
units on a scale | 34.7 (3.0) | -0.8 (4.1)
Statistical Analysis 1: Comparison: TearCare vs Warm Compress; Test type: Superiority; p < 0.0001, Simple mixed effects linear models

3. Secondary Outcome: Change in SPEED (Standard Patient Evaluation of Eye Dryness) Questionnaire Score From Baseline
Description: The Standard Patient Evaluation for Eye Dryness (SPEED) questionnaire is a well-validated instrument and widely used assessment tool for dry eye indications. The SPEED questionnaire was used to evaluate 4 symptoms (1-dryness, grittiness, or scratchiness, 2-soreness or irritation, 3-burning or watering, 3-eye fatigue) of study subjects. The maximum score is 28 (worst) and the minimum possible is 0 (best). The SPEED survey measures the severity (0-4 scale - each symptom) and frequency (0-3 scale - each symptom) of these DED symptoms. The SPEED score was calculated by adding the total of the frequency and severity scores; a score of greater than or equal to 6 may be an indicator of DED. The reported value is the mean of the change for all subjects. A negative result indicates improvement.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare | Warm Compress
Number analyzed (Participants) | 12 | 12
units on a scale | -7.9 (4.3) | -1.8 (3.6)
Statistical Analysis 1: Comparison: TearCare vs Warm Compress; Test type: Superiority; p < 0.0001, Simple mixed effects linear models

4. Secondary Outcome: Mean Change in OSDI Score From Baseline to Month 1
Description: The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire that assesses symptoms of ocular irritation associated with dry eye and the impact of these on vision-related activities. The OSDI score ranges from 0 (best possible) to 100 (worst possible). The change in OSDI questionnaire from baseline to Month 1 is the difference between the scores at the two timepoints. A negative value would indicate improvement and a positive value, a worsening. The reported value is the mean of the change for all subjects.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare | Warm Compress
Number analyzed (Participants) | 12 | 12
units on a scale | -25.3 (17.9) | -8.4 (17.1)
Statistical Analysis 1: Comparison: TearCare vs Warm Compress; Test type: Superiority; p < 0.0001, Simple mixed effects linear models

5. Secondary Outcome: Mean Change in SANDE ( Symptom Assessment in Dry Eye) Questionnaire Score From Baseline to Month 1
Description: The SANDE instrument is a simple 2-item questionnaire, that focuses on the frequency and the severity of dry eye symptoms with each measured along a visual analog scale. SANDE, because of its simplicity, is often used in routine clinical practice. For the core questions, the frequency and severity scores are multiplied together, and the square root is taken to produce an overall SANDE score from 0 (best possible) to 100 (worst possible). The mean change from baseline to month 1 is the difference in the two scores. A negative result indicates improvement.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare | Warm Compress
Number analyzed (Participants) | 12 | 12
units on a scale | -24.6 (30.9) | 2.8 (14.2)
Statistical Analysis 1: Comparison: TearCare vs Warm Compress; Test type: Superiority; p < 0.0001, Simple mixed effects linear models

ADVERSE EVENTS:
Time Frame: 6 Month
Groups:
- TearCare: Subjects will receive a 12-minute treatment session with the TearCare System followed by manual expression of the meibomian glands. This procedure will be performed at the Baseline visit. At the completion of the first 6 months, subjects will be given the option of extending their participation in the study. If they participate in the study extension, they will have the procedure performed again at the first study extension visit.
  TearCare
Arm/Group | TearCare | Warm Compress
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03006978/Prot_SAP_000.pdf